CLINICAL TRIAL: NCT03021616
Title: Evaluation of Energy Drink Consumption on Electrocardiographic, Vascular and Hematologic Parameters in Young Healthy Volunteers: A Randomized, Double Blind, Active-Controlled, Crossover Study
Brief Title: Evaluation of Energy Drinks on Electrocardiographic, Vascular and Hematologic Parameters in Healthy Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from sister study at University of the Pacific were conclusive.
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: FDG20160019H
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases
Keywords: energy drink; qtc interval; clotting time; thorough qt study
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Energy Drinks; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Energy drink (Experimental): Two 16 oz bottles of energy drink will be consumed at baseline.
  Interventions: Other: energy drink
- Moxifloxacin control (Active Comparator): 32oz of active control drink will contain 400mg moxifloxacin with inactive flavoring ingredients.
  Interventions: Other: Moxifloxacin 400mg
- placebo control (Placebo Comparator): 32oz placebo control drink
  Interventions: Other: Placebo

INTERVENTIONS:
Other: energy drink — 32oz of commercially available energy drink
  Arms: Energy drink
Other: Moxifloxacin 400mg — 400mg moxifloxacin active control drink
  Other Names: active control
  Arms: Moxifloxacin control
Other: Placebo — Placebo drink
  Arms: placebo control

SUMMARY:
This study will determine the cardiovascular effects of energy drink consumption in healthy individuals through electrocardiogram (ECG), central blood pressure assessment, and ROTEM® analysis.

DETAILED DESCRIPTION:
This is a randomized, double blind, controlled, crossover study evaluating the electrocardiographic, blood pressure, and hematological effects of an energy drink.

* Subjects who have contacted the PI/AI/SC for consideration of participation in this study will be scheduled a time to come to the Clinical Investigation Facility (CIF) Interview Room, which is a private room located on the David Grant Medical Center campus, for an initial evaluation for inclusion eligibility determination.
* At the initial evaluation subjects will be informed about the details of the study, be presented with the Informed Consent Document (ICD) and HIPAA documents and be asked to sign the appropriate forms voluntarily if they want to be a part of this study. Once consented, subjects will then be asked a series of questions to see if they qualify for inclusion in the study. A baseline ECG, Chem 7, and a peripheral blood pressure will be obtained to rule out everything but normal sinus rhythm, normal potassium level, and blood pressure less than 140/90. A cardiologist will approve every baseline ECG to allow the participant to enroll in the study.
* If the subject meets inclusion criteria and are approved by the cardiologist, they will be enrolled, and allocated a randomized participant ID number. They will also be given the "Participant Instruction Sheet".
* Participants will be asked to document their normal baseline caffeine consumption on the initial questionnaire.
* Participants will randomly be assigned to consume either two-16 oz. containers of Monster Energy® drink, original flavor, two-16 oz. containers of an active control drink, or two 16 oz. containers of a placebo drink during their first day of treatment.
* The blinding and randomization will be performed by a member of the pharmacy staff who will have the randomization code in a sealed envelope in the pharmacy. The PI, AIs and SC will be blinded. In the event of a medical emergency, unblinding a particular subject may occur upon request to the pharmacy staff from an investigator or study coordinator. Only the requested subject will be unblinded.
* The control drinks will comprise an equivalent volume. The active control drink 16 oz. bottle will contain: 200 mg moxifloxacin (dissolved tablet), carbonated water, reconstituted lime juice (readily available from supermarkets), and cherry flavoring (regularly used flavoring in compounding). The placebo drink will be the same except it will not contain moxifloxacin.
* The energy drink and control drinks will be repackaged by a member of the pharmacy staff in identical 16 oz. bottles and checked by another staff member. The active and control drinks will be made at least 24 hours but no more than 7 days in advance and will be stored in a refrigerator in a designated area within the inpatient pharmacy. Study drinks will be available for the investigator/coordinator for distribution to the participants.
* Participants will be informed on the "Participant Instruction Sheet" to refrain from caffeine or energy drink consumption for 48 hours prior to study days 1, 8, and 15. They will need to have similar work shifts 48 hours before each study day (i.e. day or night shift). In addition, participants will be instructed to be in the fasting state (no food or drink other than water) for 12 hours prior to study days 1, 8, and 15.
* On day 1, a baseline ECG, HR, peripheral and central blood pressures, and lab draw will be obtained prior to consumption of the assigned study drink. The lab draw will be used to determine baseline clotting time using ROTEM® analysis. After completion of baseline readings, subjects will have 45 minutes to consume two-16 oz. containers of Monster Energy® or either control drink as assigned. The time clock for study duration will start when the participant is issued their study drink. Repeat measurements of ECG, HR, peripheral and central blood pressures will be performed at 1, 2, 4, and 6 hours. In addition, a second lab draw will be taken at 2 hours and submitted for ROTEM® analysis to determine clotting time. At 2 hours the subject will also be provided a study-controlled breakfast. During each measurement session, participants will also be asked to "describe any adverse effects you may be experiencing". All measurements taken and responses from participants will be annotated on the participant treatment form.
* Participants may eat after lunch between hours four and five after the energy drink was consumed. They will be asked to eat approximately the same meals for lunch on the 3 study days. They may not consume additional caffeine or energy drinks not provided by the study group until after the measurements are taken 6 hours later.
* A minimum 6-day wash-out period must elapse prior to initiation of the second phase of the study, at which time the same treatment/monitoring process will occur (i.e. Day 8 or after). It will again be repeated on day 15 or after.
* Measurements will include: ECG, BP, lab draw, and questions about side effects each participant may be experiencing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female, active duty military service members or DoD beneficiaries, who are eligible to receive care at DGMC.
* Ages 18-40 years old.
* Participants must be willing to refrain from caffeine and energy drink use 48 hours prior to study days 1, 8, and 15

Exclusion Criteria:

* In an effort to recruit subjects in general good health, those with the following medical conditions or disease states will be excluded from enrollment:

  * Cardiovascular risk factors: Heart rhythm other than normal sinus, history of atrial or ventricular arrhythmia, family history of premature sudden cardiac death before the age of 60, left ventricular hypertrophy, acute myocardial ischemia, atherosclerosis, hypertension, palpitations, T-wave abnormalities, baseline corrected QT (QTc) interval greater than 440 milliseconds(ms). This will be determined on the ECG obtained during initial screening appointment, and reviewed by cardiologist and through the questionnaire responses of the participant.
  * Blood pressure at initial screening appointment or at baseline on study Day 1 greater than 140/90
  * Hypokalemia or liver abnormalities (AST/ALT abnormality) identified at initial appointment when baseline lab values will be drawn.
  * Presence of any known medical condition, confirmed through participant interview up to the discretion of the research team. Examples of these are:
* Hypertension
* Thyroid disease
* Type 1 or 2 diabetes mellitus
* Recurrent headaches
* Depression, currently receiving treatment (due to possible drug interactions)
* Any psychiatric condition or neurological disorder including seizures
* History of alcohol or drug abuse in the previous 5 years
* Ever been diagnosed or told they have or had renal or hepatic dysfunction

  * Concurrent use of ANY medication taken in an amount greater than twice a week, to include herbal products or supplements, NOT TO INCLUDE hormonal contraceptives. If less than or equal to 2 days per week, the investigator will determine if the subject is to be included or excluded based on the available literature for that medication.
  * Pregnant or lactating females will be excluded from participation with urine dipstick tests used to confirm pregnancy (pregnancy test performed before each treatment session, days 1, 8 and 15)
  * All non-English speaking / writing subjects and those that do not understand the study or consent process will be excluded from the study due to unavailability of medical qualified translator at all times during the study.
  * If the subject refuses to sign the informed consent document or HIPAA Authorization, they will be excluded as well.
  * Allergy to any substance in the study design.
  * Any other medical reason that at the discretion of the investigators would pose a risk to the health of the subject.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
QTc interval change from baseline in each of 3 arms | 1 hour post consumption
Central systolic blood pressure change from baseline in each of 3 arms | 1 hour post consumption
Peripheral systolic blood pressure change from baseline in each of 3 arms | 1 hour post consumption
QTc interval change from baseline in each of 3 arms | 2 hours post consumption
QTc interval change from baseline in each of 3 arms | 4 hours post consumption
QTc interval change from baseline in each of 3 arms | 6 hours post consumption
central systolic blood pressure change from baseline in each of 3 arms | 2 hours post consumption
central systolic blood pressure change from baseline in each of 3 arms | 4 hours post consumption
central systolic blood pressure change from baseline in each of 3 arms | 6 hours post consumption
Peripheral systolic blood pressure change from baseline in each of 3 arms | 2 hours post consumption
Peripheral systolic blood pressure change from baseline in each of 3 arms | 4 hours post consumption
Peripheral systolic blood pressure change from baseline in each of 3 arms | 6 hours post consumption

SECONDARY OUTCOMES:
Thromboelastometry changes from baseline in each of 3 arms | 2 hours post consumption
ECG parameter changes from baseline in each of 3 arms | 1 hour post consumption
ECG parameter changes from baseline in each of 3 arms | 2 hours post consumption
ECG parameter changes from baseline in each of 3 arms | 4 hours post consumption
ECG parameter changes from baseline in each of 3 arms | 6 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kelly, PharmD, Principal Investigator — David Grant Medical Center
Locations (1):
- David Grant Medical Center, Travis Air Force Base, California, United States

REFERENCES:
- [Background] Ammar R, Song JC, Kluger J, White CM. Evaluation of electrocardiographic and hemodynamic effects of caffeine with acute dosing in healthy volunteers. Pharmacotherapy. 2001 Apr;21(4):437-42. doi: 10.1592/phco.21.5.437.34502. PMID 11310517
- [Background] Biewenga J, Keung C, Solanki B, Natarajan J, Leitz G, Deleu S, Soons P. Absence of QTc Prolongation with Domperidone: A Randomized, Double-Blind, Placebo- and Positive-Controlled Thorough QT/QTc Study in Healthy Volunteers. Clin Pharmacol Drug Dev. 2015 Jan;4(1):41-48. doi: 10.1002/cpdd.126. Epub 2014 May 30. PMID 26097791
- [Background] Carlson GF, Tou CK, Parikh S, Birmingham BK, Butler K. Evaluation of the effect of dapagliflozin on cardiac repolarization: a thorough QT/QTc study. Diabetes Ther. 2011 Sep;2(3):123-32. doi: 10.1007/s13300-011-0003-2. Epub 2011 Jun 24. PMID 22127822
- [Background] Cassella JV, Spyker DA, Yeung PP. A randomized, placebo-controlled repeat-dose thorough QT study of inhaled loxapine in healthy volunteers. Int J Clin Pharmacol Ther. 2015 Nov;53(11):963-71. doi: 10.5414/CP202457. PMID 26501204
- [Background] Elitok A, Oz F, Panc C, Sarikaya R, Sezikli S, Pala Y, Bugan OS, Ates M, Parildar H, Ayaz MB, Atici A, Oflaz H. Acute effects of Red Bull energy drink on ventricular repolarization in healthy young volunteers: a prospective study. Anatol J Cardiol. 2015 Nov;15(11):919-22. doi: 10.5152/akd.2015.5791. Epub 2015 Mar 5. PMID 25868042
- [Background] Furie B, Furie BC. Mechanisms of thrombus formation. N Engl J Med. 2008 Aug 28;359(9):938-49. doi: 10.1056/NEJMra0801082. No abstract available. PMID 18753650
- [Background] Hajsadeghi S, Mohammadpour F, Manteghi MJ, Kordshakeri K, Tokazebani M, Rahmani E, Hassanzadeh M. Effects of energy drinks on blood pressure, heart rate, and electrocardiographic parameters: An experimental study on healthy young adults. Anatol J Cardiol. 2016 Feb;16(2):94-9. doi: 10.5152/akd.2015.5930. Epub 2015 Mar 23. PMID 26467367
- [Background] Litwin JS, Benedict MS, Thorn MD, Lawrence LE, Cammarata SK, Sun E. A thorough QT study to evaluate the effects of therapeutic and supratherapeutic doses of delafloxacin on cardiac repolarization. Antimicrob Agents Chemother. 2015;59(6):3469-73. doi: 10.1128/AAC.04813-14. Epub 2015 Apr 6. PMID 25845864
- [Background] Kumagai Y, Hasunuma T, Sakai S, Ochiai H, Samukawa Y. Randomized, Controlled, Thorough QT/QTc Study Shows Absence of QT Prolongation with Luseogliflozin in Healthy Japanese Subjects. PLoS One. 2015 Oct 7;10(10):e0139873. doi: 10.1371/journal.pone.0139873. eCollection 2015. PMID 26444986
- [Background] Malinauskas BM, Aeby VG, Overton RF, Carpenter-Aeby T, Barber-Heidal K. A survey of energy drink consumption patterns among college students. Nutr J. 2007 Oct 31;6:35. doi: 10.1186/1475-2891-6-35. PMID 17974021
- [Background] Myers MG. Effect of caffeine on blood pressure beyond the laboratory. Hypertension. 2004 Apr;43(4):724-5. doi: 10.1161/01.HYP.0000120970.49340.33. Epub 2004 Feb 16. No abstract available. PMID 14967826
- [Background] Ohno Y, Kanno Y, Takenaka T. Central blood pressure and chronic kidney disease. World J Nephrol. 2016 Jan 6;5(1):90-100. doi: 10.5527/wjn.v5.i1.90. PMID 26788468
- [Background] Phan JK, Shah SA. Effect of caffeinated versus noncaffeinated energy drinks on central blood pressures. Pharmacotherapy. 2014 Jun;34(6):555-60. doi: 10.1002/phar.1419. Epub 2014 Mar 19. PMID 24644139
- [Background] Pommerening MJ, Cardenas JC, Radwan ZA, Wade CE, Holcomb JB, Cotton BA. Hypercoagulability after energy drink consumption. J Surg Res. 2015 Dec;199(2):635-40. doi: 10.1016/j.jss.2015.06.027. Epub 2015 Jun 18. PMID 26188956
- [Background] Seifert SM, Schaechter JL, Hershorin ER, Lipshultz SE. Health effects of energy drinks on children, adolescents, and young adults. Pediatrics. 2011 Mar;127(3):511-28. doi: 10.1542/peds.2009-3592. Epub 2011 Feb 14. PMID 21321035
- [Background] Shah SA, Occiano A, Nguyen TA, Chan A, Sky JC, Bhattacharyya M, O'Dell KM, Shek A, Nguyen NN. Electrocardiographic and blood pressure effects of energy drinks and Panax ginseng in healthy volunteers: A randomized clinical trial. Int J Cardiol. 2016 Sep 1;218:318-323. doi: 10.1016/j.ijcard.2016.05.007. Epub 2016 May 13. PMID 27240158
- [Background] Shah SA, Chu BW, Lacey CS, Riddock IC, Lee M, Dargush AE. Impact of Acute Energy Drink Consumption on Blood Pressure Parameters: A Meta-analysis. Ann Pharmacother. 2016 Oct;50(10):808-15. doi: 10.1177/1060028016656433. Epub 2016 Jun 23. PMID 27340146